CLINICAL TRIAL: NCT04780555
Title: Evaluation of Pain Symptoms Correlation With Biochemical and Radiological Findings in COVID-19
Brief Title: Evaluation of Musculoskeletal System Symptoms and Biochemical Parameters in COVID-19
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Elif yaksi, Medical Doctor, Abant Izzet Baysal University
Other Study IDs: AIBU-FTR-EY-02
Record Dates: First submitted 2021-02-21; First posted 2021-03-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Covid19
Keywords: pain
MeSH Terms: conditions — COVID-19; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral venous blood specimens will be collected using standard surgical procedures during presentation and were investigated in the Abant İzzet Baysal University Medical Faculty central laboratory. Complete blood count parameters (hemoglobin, leukocytes, erythrocytes, platelets, and leukocyte subtypes) will be analyzed using a Syxmex XN-1000 (Kobe, Japan) automatic analyzer. D-dimer and fibrinogen parameters will be measured on a Sysmex CS-2500 (Kobe, Japan) device, and biochemical parameters (CRP, ferritin, procalcitonin, LDH, troponin) on an automatic biochemical analyzer (Abbott Architect C8000, USA). In addition, the NLR will be calculated by dividing the absolute neutrophil count by the absolute lymphocyte count.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The neutrophil-lymphocyte ratio (NLR) used to demonstrate inflammatory status in recent years can be calculated by dividing the absolute neutrophil count by the absolute lymphocyte count at routine blood tests.

DETAILED DESCRIPTION:
Dysregulation in immune responses has been reported in association with hyperinflammation in COVID-19 patients, NLR has been linked to the severity of the patient's clinical status, and an increase in NLR is reported to be an independent risk factor for in-hospital mortality. Pain is a frequently seen symptom at the onset of viral infections and throughout the course of the disease. Although the pain mechanisms triggered by viral pathogens are not yet entirely understood, pain is thought to arise as a result of direct activation of nociceptor neurons by pathogens and their interaction with molecular ligands. Toll-like receptor 7 (TLR7), a pathogen recognition receptor that plays an important role in immune responses to viruses by binding to viral RNA, is known to be involved in pain development in different RNA virus infections. Park et al. showed that extracellular micro RNAs activate nociceptive neurons via the TLR7 pathway. Although these mechanisms have been demonstrated for different viral infections, the viral pathogenesis leading to pain in COVID-19 is still unclear. The purpose of this study was to investigate the prevalence of headache and muscular pain in patients diagnosed with COVID-19 and to determine the relationship between these symptoms and inflammatory parameters.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70
* Diagnosed with COVID-19

Exclusion Criteria:

* Patients with suspected SARS-CoV-2 infection, with two negative RT-PCR tests, hospitalized in the intensive care unit during inclusion in the study
* Musculoskeletal pains in the previous three months, with diseases capable of causing myalgia prior to diagnosis (such as fibromyalgia and inflammatory muscle disease)
* Cognitive disorders capable of preventing history-taking and physical examination such as mental disability and dementia,
* previous history of headache (migraine, tension type headache)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-65 and diagnosed with COVID-19 will be included in the study.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-07-25 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Neutrophil-lymphocyte ratio (NLR) | Baseline
  It can be calculated by dividing the absolute neutrophil count by the absolute lymphocyte count at routine blood tests
D-dimer | Baseline
  Peripheral venous blood specimens were collected using standard surgical procedures
Fibrinogen | Baseline
  Peripheral venous blood specimens were collected using standard surgical procedures

CONTACTS AND LOCATIONS:
Overall Officials: Nalan Doğan, MD, Principal Investigator — Beykoz State Hospital; Dursun Karakaş, MD, Principal Investigator — Sancaktepe Şehit İlhan Varank Research Hospital; Osman Yakşi, MD, Principal Investigator — Abant İzzet Baysal University Medical Faculty
Locations (1):
- Elif Yakşi, Merkez, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No